CLINICAL TRIAL: NCT03340051
Title: Episodic Thinking (ET) as a Candidate Technique to Reduce Alcohol Consumption
Brief Title: Remote Alcohol Monitoring and Episodic Thinking
Acronym: RMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Stephen LaConte, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMET/15-955
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Dependence; Alcohol-Related Disorders
MeSH Terms: conditions — Alcoholism; Alcohol-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFT group (Active Comparator): Episodic Future Thinking (EFT) is the intervention in this arm. EFT participants will generate positive future events they are looking forward to and that could happen at different future time points (e.g., in 2 weeks, 1 month, 6 months, 1 year). Participants will be instructed to use and think about their episodic cues as they make decisions.
  Interventions: Behavioral: Episodic Future Thinking (EFT)
- ERT group (Placebo Comparator): Episodic Recent Thinking (ERT) is the intervention in this arm. ERT participants will list positive recent events (events that have already happened) that they enjoyed that occurred at different past time points (e.g., 12 hours ago, 24 hours ago, a week ago). Participants will be instructed to use and think about their episodic cues as they make decisions.
  Interventions: Behavioral: Episodic Recent Thinking (ERT)

INTERVENTIONS:
Behavioral: Episodic Future Thinking (EFT) — EFT participants will generate positive future events they are looking forward to and that could happen at different future time points (e.g., in 2 weeks, 1 month, 6 months, 1 year). Participants will be instructed to use and think about their episodic cues as they make decisions.
  Arms: EFT group
Behavioral: Episodic Recent Thinking (ERT) — ERT participants will list positive recent events (events that have already happened) that they enjoyed that occurred at different past time points (e.g., 12 hours ago, 24 hours ago, a week ago). Participants will be instructed to use and think about their episodic cues as they make decisions.
  Arms: ERT group

SUMMARY:
Nearly 18% of United States adults meet criteria for alcohol dependence sometime in their lifetime, with only 24% of those individuals ever receiving any treatment for their disorder (Hasin et al., 2007). The pervasiveness of alcohol dependence indicates a need for continued development of high-impact treatments that are both effective and easily disseminated to a broad population. Recent evidence indicates that Episodic Future Thinking (EFT), the ability to self-project and pre-experience a future event, can help individuals to make changes to habitual behaviors, such as alcohol drinking (Snider et al., 2016). In this study, the investigators will evaluate the efficacy of EFT to help individuals reduce alcohol consumption. The investigators anticipate that EFT will result in a reduction in alcohol consumption over a 2-week experimental period when compared to the control group.

DETAILED DESCRIPTION:
After the initial consent and assessment sessions, participants will be asked to provide daily self-report assessments of previous-day drinking over cell phone for 7 days with no other study intervention taking place. The purpose for this baseline period is to quantify baseline drinking patterns and ensure that the participant reliably responds to and conveys study information via cell phone. At the end of this baseline period, participants who indicated adaquate patterns of drinking and successfully reported their level of drinking will be invited to continue in the study. Participants will return to the laboratory to be provided with a SOBERLINK breathalyzer and be given instruction in its use. The SOBERLINK device will automatically upload breathalyzer results, the participant's location, and the picture of the user to a centralized, secure website where the data will be available to research staff.

Participants will be counterbalanced to either the active or control group based on alcohol use (e.g., average drinks per day). Both groups will be exposed to the same treatment events. The intervention period will last for 14 consecutive days, with three breathalyzer screens per day. During this 14-day period as they did during the baseline period, participants will self-report their previous-day alcohol use daily with a text message and/or phone call. Assessment sessions will be conducted prior to the intervention, immediately following the intervention, and at a 1-month follow-up.

All participants will either be allowed to use their own personal cell phone for study communications or receive a prepaid cell phone with service through a nationwide cell phone service provider. The study-provided phones include usage controls, allowing us to restrict phone communication to a study phone and 911 service.

Throughout the intervention phase of the experiment, participants will be required to submit three daily breathalyzer assessments at the predetermined times. They will be reminded via text message when a sample is to be collected, and samples will be accepted up to 15 minutes before the scheduled time and 30-60 minutes after the scheduled time, giving the participant 45-75 minutes total to submit the sample.

Participants will be assigned to either the active Episodic Future Thinking (EFT) condition or the control Episodic Recent Thinking (ERT) condition. EFT participants will generate positive future events they are looking forward to and that could happen at different future time points (e.g., in 2 weeks, 1 month, 6 months, 1 year) and participants in the ERT condition will list positive recent events (events that have already happened) that they enjoyed that occurred at different past time points (e.g., 12 hours ago, 24 hours ago,1 week ago). Participants will be instructed to use and think about their episodic cues as they make decisions. All participants will be provided with a copy of their episodic cues to take home with them and will receive periodic text messages from research staff to remind them of their cues. In addition, each day, participants will be asked to report how many alcoholic drinks they consumed the previous day (from the time they awoke to the time they fell asleep). Participants will be allowed to report this information via text message or phone call. Participants will receive a reminder to report their previous-day drinking with text messages, followed by a phone call if they haven't contacted us by early evening.

Assessment sessions will be completed before the 14-day intervention period, immediately after the 14-day intervention period, and at a 1-month follow-up. Participants will complete a battery of questionnaires and tasks grouped into three general categories: measures of substance use (including a urine test for drug use and a breath sample to test for recent alcohol use), clinically relevant measures including treatment acceptability, and measures of alcohol value and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. provide written informed consent
2. be 18-65 years old
3. meet DSM-V criteria for moderate or severe alcohol use disorder
4. express a desire to quit or cut down on their drinking.

Exclusion Criteria:

Individuals who are:

1. pregnant or lactating
2. meet DSM-V criteria for any other moderate or severe substance use disorders (excluding caffeine, nicotine, and marijuana),
3. score 23 or greater on the Alcohol Withdrawal Symptom Checklist (a score indicating that medication would be likely required to manage alcohol detoxification)
4. use prescribed or over-the-counter medicines containing alcohol
5. participated in any previous studies that included EFT at the Addiction Recovery Research Center in the last three months
6. have immediate plans to move out of the area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Change in average daily alcohol consumption | Self report of daily alcohol use will be collected every morning for 7 days after the first session (baseline measure) and for 14 days after the second session and the averages of the 7- and 14-day periods will be compared (pre-post intervention).
  Change in average daily alcohol consumption collected using self reports

SECONDARY OUTCOMES:
Change in delay discounting rate | At the first session (baseline measures), third session (after 3 weeks/post-intervention), and the 1 month follow up assessments. The average discounting rates within each group will be compared pre-post intervention
  Discounting rates will be measured using adjusting amount delay discounting and minute delay discounting tasks
Change in intensity of alcohol demand | At the first session (baseline measures), third (after 3 weeks/post-intervention), and the 1 month follow up assessments. The average scores within each group will be compared pre-post intervention
  Change in intensity of alcohol demand will be determined from an alcohol demand curve generated via an Alcohol Purchase Task (APT)
Change in elasticity of alcohol demand | At the first session (baseline measures), third (after 3 weeks/post-intervention), and the 1 month follow up assessments. The average scores within each group will be compared pre-post intervention
  Change in elasticity of alcohol demand will be determined from an alcohol demand curve generated via an Alcohol Purchase Task (APT)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, PhD, Principal Investigator — Virginia Tech Carilion School of Medicine and Research Institute
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Athamneh LN, Brown J, Stein JS, Gatchalian KM, LaConte SM, Bickel WK. Future thinking to decrease real-world drinking in alcohol use disorder: Repairing reinforcer pathology in a randomized proof-of-concept trial. Exp Clin Psychopharmacol. 2022 Jun;30(3):326-337. doi: 10.1037/pha0000460. Epub 2021 Apr 22. PMID 35041442

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03340051/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03340051/SAP_001.pdf